CLINICAL TRIAL: NCT04348409
Title: Proof of Concept, Multicentre, Parallel, Randomized, Double-blind Clinical Trial to Assess the Safety and Efficacy of Nitazoxanide 600 mg Compared to Placebo in the Treatment of Hospitalized Patients With COVID-19 in Moderate Condition.
Brief Title: Efficacy and Safety of Nitazoxanide for the Treatment of Hospitalized Patients With Moderate COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: Farmoquimica S.A. (Industry); Hospital Vera Cruz (Other); Hospital Casa de Saúde - Vera Cruz - Campinas - SP - Brazil (Unknown); Centro de Genomas - UNIFESP (Unknown); Emilio Ribas Institute of Infectious Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NITFQM0320OR
Record Dates: First submitted 2020-04-03; First posted 2020-04-16 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either nitazoxanide or placebo (1:1).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nitazoxanide (Experimental): Patients will receive nitazoxanide 600 mg BID for 7 days.
  Interventions: Drug: Nitazoxanide Tablets
- Placebo (Placebo Comparator): Patients will receive placebo BID for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide Tablets — Patients will receive nitazoxanide 600 mg BID for 7 days
  Arms: nitazoxanide
Drug: Placebo — Patients will receive placebo BID for 7 days
  Arms: Placebo

SUMMARY:
This is a proof of concept study to evaluate the efficacy of nitazoxanide (600 mg BID) to treat hospitalized patients with moderate COVID-19.

DETAILED DESCRIPTION:
This is a proof of concept study to evaluate the efficacy of nitazoxanide (600 mg BID) to treat hospitalized patients with moderate COVID-19.

The aim is to demonstrate a decrease in hospital related complications among patients who are hospitalized with moderate COVID-19 by treating them with nitazoxanide for 7 days on top of standard care compared to patients who receive standard care and placebo.

Patients hospitalized with confirmed diagnosis of COVID-19 will be randomized to receive either nitazoxanide or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from patient or legal representative.
2. Male or female, aged ≥ 18 years;
3. Laboratory confirmation of 2019-nCoV infection by reverse-transcription polymerase chain reaction (RT-PCR) from any diagnostic sampling source;
4. Signs of respiratory failure requiring oxygen therapy
5. Hospitalized for up to 36h with non-invasive ventilation
6. Negative result for pregnancy test (if applicable).

Exclusion Criteria:

1. Participating in another RCT in the past 12 months;
2. Known allergy to nitazoxanide
3. Severely reduced LV function;
4. Severely reduced renal function;
5. Pregnancy or breast feeding;
6. Use of hydroxychloroquine and/or azithromycin in the past 15 days;
7. Any other clinical condition which, in the opinion of the principal investigator, would not allow safe completion of the protocol and safe administration of the investigational products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Viral load | day 1, 4, 7, 14 and 21
  PCR will be done to evaluate the change in viral load

SECONDARY OUTCOMES:
Evolution of acute respiratory syndrome | 21 days
  Time to wean off oxygen supplementation
Change in Clinical Condition | 21 days
  WHO Ordinal Scale for Clinical Improvement that measures illness severity over time (0=uninfected; ambulatory, no limitation of activities=1; ambulatory, limitation of activities=2, hospitalized no oxygen therapy=3; hospitalized oxygen by mask or nasal prongs=4; hospitalized non invasive ventilation or high-flow oxygen=5; hospitalized intubation or mechanical ventilation=6; hospitalized ventilation + additional organ support=7; death=8)
Hospital discharge | 21 days
  Time to be discharged from hospital
Rate of mortality within 21-days | 21 days
  Evaluation of change in acute respiratory syndrome
Need of mechanical ventilation | 21 days
  Evaluation of change in acute respiratory syndrome

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Hospital Vera Cruz, Campinas, São Paulo
  - Centro de Genomas, São Paulo
  - Hospital Emílio Ribas, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.

REFERENCES:
- [Derived] Blum VF, Cimerman S, Hunter JR, Tierno P, Lacerda A, Soeiro A, Cardoso F, Bellei NC, Maricato J, Mantovani N, Vassao M, Dias D, Galinskas J, Janini LMR, Santos-Oliveira JR, Da-Cruz AM, Diaz RS. Nitazoxanide superiority to placebo to treat moderate COVID-19 - A Pilot prove of concept randomized double-blind clinical trial. EClinicalMedicine. 2021 Jul;37:100981. doi: 10.1016/j.eclinm.2021.100981. Epub 2021 Jun 27. PMID 34222847